CLINICAL TRIAL: NCT00110331
Title: Central Nervous System Disease in HIV-infected Children on HAART
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050150; 05-C-0150
Record Dates: First submitted 2005-05-05; First posted 2005-05-06 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2014-09-09

CONDITIONS: HIV Infections; Central Nervous System Diseases
Keywords: Encephalopathy; Neuroimaging; Cognition; Neuroinflammation; Opportunistic Infections; HIV; Central Nervous System Disease; Bipolar Disorder; Attention Deficit Hyperactivity Disorder; ADHD; Major Depression; Psychosis
MeSH Terms: conditions — HIV Infections; Central Nervous System Diseases; Brain Diseases; Neuroinflammatory Diseases; Opportunistic Infections; Bipolar Disorder; Attention Deficit Disorder with Hyperactivity; Depressive Disorder, Major; Psychotic Disorders

SUMMARY:
This study will examine how HIV affects the brain and nervous system, learning, and behavior in children on highly active antiretroviral therapy (HAART). Although HAART has resulted in fewer HIV-infected children getting sick and even fewer dying from AIDS, many children on this treatment regimen develop significant brain or nervous system problems, such as learning difficulties, attention problems, hyperactivity, and depression.

People who acquired HIV disease in the first decade of life and who have evidence of central nervous system (CNS) disease (e.g., encephalopathy, CNS compromise, ADHD, bipolar disease, major depression or psychosis) may be eligible for this study. Candidates are screened with a medical history, physical examination, neuropsychological testing and a CT scan of the head, if one has not been done within 12 months of entering the study.

Participants undergo the following tests and procedures:

* MRI and MRS scan of the head: These tests use a magnetic field and radio waves to obtain images of the brain and detect changes in certain brain chemicals that may be affected by HIV infection. Both procedures are done at the same time. The patient lies on a table that is moved into the scanner (a narrow cylinder), wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. The procedure lasts about 50 to 60 minutes, during which time the patient can communicate with the staff.
* Neuropsychological testing: Patients' thinking and behavior are evaluated with tests to measure their memory, attention, language, problem-solving, academic, and motor skills and questionnaires to assess behavioral and emotional functioning, quality of life, and adherence to HIV medication. Parents are also asked to complete questionnaires assessing their child's behavioral and emotional functioning, quality of life, important life events, and adherence to HIV medication.
* Lumbar puncture (spinal tap): Cerebrospinal fluid (CSF) is collected for analysis. For this procedure, a local anesthetic is given and a needle is inserted in the space between the bones in the lower back where the CSF circulates below the spinal cord. Some fluid is collected through the needle. Blood tests and a physical examination are done before the procedure to make sure it can be done as safely as possible. Patients may also be sedated to prevent any discomfort.
* Follow-up: The blood tests, MRI and MRS scans and spinal tap are repeated 1 and 2 years after the initial evaluation.

Some blood and spinal fluid samples from participants are stored for possible future studies related to HIV research

DETAILED DESCRIPTION:
Background:

Highly active antiretroviral therapy (HAART) has altered the natural history of HIV disease in children.

A significant minority of HIV-infected children has evidence of ongoing CNS disease.

Specific markers for CNS disease, factors predictive of risk for neurological decline, and pathophysiologic mechanisms have not yet been identified in HIV-infected children.

Objective:

To explore the clinical features (neurological and psychiatric exams, neuropsychological evaluation, and neuroimaging), viral and neuroinflammatory factors, anatomic changes (brain MRI) and patterns of brain metabolites (1H-MRS) associated with HIV-related CNS disease in HIV-infected children in the HAART era.

Eligibility:

HIV disease acquired in the first decade of life.

Evidence of CNS disease (classification of encephalopathy or CNS compromise or diagnosis of ADHD, bipolar disease, major depression, or psychosis).

Design:

Serial neurologic and psychiatric examinations, neuropsychologic test, neuroimaging, and CSF sampling will be performed once a year for a total of 3 evaluations.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. HIV disease acquired in the first decade of life.
2. Evidence of CNS disease (at least one of the following):

   * Classification of encephalopathy or CNS compromise.
   * Diagnosis of ADHD, bipolar disease, major depression, or psychosis
3. For children greater than 7 years, ability to give assent if developmentally appropriate.

EXCLUSION CRITERIA:

1. Inability or unwillingness to provide informed consent for subjects greater than 18 years, and inability or unwillingness of one parent / legal guardian to provide consent for subjects less than 18 years.
2. Clinically significant, unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction) which in the judgment of the Principal Investigator or Chairpersons would compromise the patient's ability to tolerate this study or is likely to interfere with the study procedures or results

Lumbar Puncture Exclusion Criteria:

1. Increased intracranial pressure (head imaging and neurologic examination to be performed prior to LP)
2. Spinal cord lesion (to be screened by neurologic examination; spine imaging if clinically indicated)
3. Platelet count less than 75,000/mm(3)
4. Abnormal PT/PTT
5. Focal suppuration at puncture site

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2005-05-03; Study Completion 2014-09-09

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Hazra, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gortmaker SL, Hughes M, Cervia J, Brady M, Johnson GM, Seage GR 3rd, Song LY, Dankner WM, Oleske JM; Pediatric AIDS Clinical Trials Group Protocol 219 Team. Effect of combination therapy including protease inhibitors on mortality among children and adolescents infected with HIV-1. N Engl J Med. 2001 Nov 22;345(21):1522-8. doi: 10.1056/NEJMoa011157. PMID 11794218
- [Background] Belman AL, Ultmann MH, Horoupian D, Novick B, Spiro AJ, Rubinstein A, Kurtzberg D, Cone-Wesson B. Neurological complications in infants and children with acquired immune deficiency syndrome. Ann Neurol. 1985 Nov;18(5):560-6. doi: 10.1002/ana.410180509. PMID 3000281
- [Background] Tamula MA, Wolters PL, Walsek C, Zeichner S, Civitello L. Cognitive decline with immunologic and virologic stability in four children with human immunodeficiency virus disease. Pediatrics. 2003 Sep;112(3 Pt 1):679-84. doi: 10.1542/peds.112.3.679. PMID 12949303